CLINICAL TRIAL: NCT05747430
Title: Randomized, Controlled, Double-Masked Study to Evaluate the Efficacy of IRX-101 in Reducing Post-Intravitreal Injection Pain and Corneal Epitheliopathy
Brief Title: SteRilizing Eye SoLution to ImprovE Patient ComFort (RELIEF)
Acronym: RELIEF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iRenix Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRX-2022-002
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to IRX-101 or Providone-Iodine
Who Masked: Participant, Investigator
Masking Description: Treatment assignment will be unknown (or masked) to the study subjects, the evaluating physician, the Sponsor and its agents (with the exception of personnel performing randomization, unmasked drug accountability study monitors, and corporate compliance staff). The treating physician will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IRX-101 (Experimental): Subjects randomized to IRX-101 will receive the investigational product, IRX-101.
  Interventions: Drug: IRX-101
- 5% Povidone-iodine (Active Comparator): Subjects randomized to this arm will receive the standard of care, Providone-iodine, at a concentration of 5%.
  Interventions: Drug: Providone-Iodine

INTERVENTIONS:
Drug: IRX-101 — IRX-101 is a novel ocular anti-septic
  Arms: IRX-101
Drug: Providone-Iodine — 5% Providone-Iodine
  Arms: 5% Povidone-iodine

SUMMARY:
This is a randomized, double-masked study to evaluate the tolerability and safety of IRX-101 versus 5% povidone-iodine (PI) in subjects receiving intravitreal anti-VEGF injections. The study will be conducted in up to 15 centers in the United States (US).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, ≥ 18 years of age and receiving intravitreal anti-VEGF injections in one or both eyes

Exclusion Criteria:

1. Current or past diagnosis of endophthalmitis
2. Current diagnosis of uveitis
3. Monocular patients (vision 20/100 or worse in one eye) who are receiving injections in the better seeing eye
4. Current use of viscous lidocaine products for ocular anesthesia prior to IVT
5. Currently receiving intravitreal steroid injections
6. Concurrent participation in another clinical trial
7. Females who are pregnant, planning to become pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Safety of new drug | 1-hour and 1-week post-treatment
  Safety will be measured via slit lamp and fundoscopic examinations

SECONDARY OUTCOMES:
Mean corneal fluorescein staining scores | Immediately following intraviteral injection
  Compare mean corneal fluorescein staining scores obtained after IVT in the IRX-101 and standard of care groups; corneal staining will be obtained using the validated Oxford Corneal Staining scale of 0 (no staining) to 5 (maximal staining)
Patient-reported post-injection pain scores | 1-hour post-administration
  Compare mean patient-reported post-injection pain scores 1-hour post-administration; pain will be assessed using the visual analog pain scale, a validated patient-reported outcome measure (questionnaire) for assessing patient's subjective pain and discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, MD, Study Chair — Founder
Locations (1):
- Edward Wood, MD, Round Rock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided